CLINICAL TRIAL: NCT00988741
Title: A Randomized Controlled Phase 2 Trial of ARQ 197 in Patients With Unresectable Hepatocellular Carcinoma (HCC) Who Have Failed One Prior Systemic Therapy
Brief Title: Trial of ARQ 197 in Patients With Unresectable Hepatocellular Carcinoma (HCC) Who Have Failed One Prior Systemic Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARQ 197-215
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Unresectable; Hepatocellular; Carcinoma
MeSH Terms: conditions — Carcinoma | interventions — ARQ 197

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARQ 197 (Experimental)
  Interventions: Drug: ARQ 197
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARQ 197 — The investigational drug ARQ 197 is supplied as capsules. A dose of 360 mg (3 capsules of 120 mg each) of ARQ 197 will be administered by mouth BID, once in the morning and once in the evening with meals, for a total daily dose of 720 mg. Under Amendment 2, a dose of 240 mg (2 capsules of 120 mg each) of ARQ 197/placebo will be administered by mouth BID, once in the morning and once in the evening with meals, for a total daily dose of 480 mg. A treatment cycle is defined as 4 weeks for both treatment arms. Cycles will be repeated every 4 weeks (28 days) based on toxicity and response.
  Other Names: Tivantinib
  Arms: ARQ 197
Drug: Placebo — The placebo is provided in a capsule form.
  Arms: placebo

SUMMARY:
This is a global randomized, placebo-controlled, double-blinded Phase 2 study designed to compare treatment of ARQ 197 versus placebo in patients with unresectable HCC who had radiographic disease progression after systemic first line therapy or were unable to tolerate the therapy.

DETAILED DESCRIPTION:
Patients will be randomly assigned in a 2:1 ratio to receive ARQ 197 or placebo. The treatment assignment will be stratified based on Eastern Cooperative Oncology Group (ECOG) performance status (PS), and vascular invasion status. The treatment with ARQ 197 or placebo will be continued until progression of disease, unacceptable toxicity, or another discontinuation criterion listed in this protocol is met.

After radiographic disease progression is documented, treatment assignment will be unblinded. Patients who were assigned to placebo arm and had documented radiographic disease progression will have the option to receive ARQ 197 and will be evaluated for objective response rate and disease control rate continuously.

The study will continue until 78 total time to progression events are reached. At the end of study, all remaining patients still on treatment will have the option to be rolled over to another study to continue their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent granted prior to initiation of any study-specific screening procedures
* 18 year of age or older
* Histologically or cytologically confirmed HCC
* Archival, fresh core needle biopsy or fine needle aspiration (FNA) tumor samples
* Received at least one cycle of prior systemic therapy (at least 3 weeks for continuously administered drugs) and experienced radiographic disease progression or was unable to tolerate therapy. If intolerance was manifested by a Grade 3 or 4 event of such nature that re-challenge is not acceptable, less than 3 weeks of continuous administration will be allowed
* Discontinued prior treatment for at least 4 weeks, or at least 2 weeks (14 days) if drug was administered continuously and orally (e.g. sorafenib or sunitinib), prior to the study randomization
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤1
* Local or loco-regional therapy (i.e., surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) must have been completed ≥4 weeks prior to randomization
* Measurable disease as defined by a modified version of the revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (see section 9). Tumor lesions previously treated with local therapy should demonstrate clear dimensional increase by radiographic assessment in order to be selected as target lesion(s) at baseline. (Radiological assessment needs to be redone within 7 days prior to randomization if the pre-study AFP level has increased by more than 30% since the last AFP level taken one to four months prior to randomization)
* Adequate bone marrow, liver, and renal functions at Pre-Study Visit, defined as:

  * Platelet count ≥ 60 × 10^9/L
  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥1.5 × 10^9/L
  * Total bilirubin ≤ 2 mg/dL
  * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 5 × upper limit of normal (ULN)
  * Serum creatinine ≤1.5 × ULN
  * International normalized ratio (INR) 0.8 to 1.4 or ≤3 for patients receiving anticoagulant such as coumadin or heparin. Patients who are therapeutically anticoagulated are allowed to participate provided that no prior evidence of underlying abnormality exists in these parameters
  * Albumin ≥ 2.8 g/dL
* Women of childbearing potential must have a negative pregnancy test performed within ten days prior to the start of study drug
* Male and female subjects of child-bearing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last investigational drug dose received

Exclusion Criteria:

* More than 1 prior systemic regimen
* Child-Pugh B-C cirrhotic status
* Previous or concurrent cancer that is distinct from HCC in primary site or histology, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated >3 years prior to enrollment is permitted
* History of congestive heart failure defined as Class II to IV per New York Heart Association (NYHA) classification within 6 months prior to study entry; active coronary artery disease (CAD); clinically significant bradycardia or other uncontrolled, cardiac arrhythmia defined as ≥Grade 3 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, or uncontrolled hypertension; myocardial infarction occurring within 6 months prior to study entry (myocardial infarction occurring >6 months prior to study entry is permitted)
* Active clinically serious infections defined as ≥ Grade 3 according to NCI CTCAE, version 4.0.
* Substance abuse, medical, psychological or social conditions that may, in the opinion of the Investigator, interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her protocol compliance
* Known human immunodeficiency virus (HIV) infection
* Pregnancy or breast-feeding
* History of liver transplant
* Inability to swallow oral medications
* Clinically significant gastrointestinal bleeding occurring ≤4 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Evaluate time to progression among all patients treated with ARQ 197 compared to placebo | Patients will be evaluated every 6 weeks until unacceptable toxicity, disease progression or another discontinuation criterion is met

SECONDARY OUTCOMES:
Evaluate progression-free survival, overall survival, objective response rate and disease control rate among all patients treated with ARQ 197 compared to placebo. | Patients will be evaluated for these endpoints every 6 weeks
Evaluate objective response rate in crossover population following radiographic disease progression on placebo. | Patients will be evaluated for these endpoints every 6 weeks
Further characterize the safety of ARQ 197 in patients with unresectable HCC | While on therapy, patients will be evaluated for safety every 4 weeks
Further evaluate pharmacokinetics of ARQ 197. | Patients will be evaluated monthly for the first 3 months

CONTACTS AND LOCATIONS:
Locations (21):
- United States (3):
  - Los Angeles, California
  - Tampa, Florida
  - Galveston, Texas
- Belgium (2):
  - Brussels
  - Ghent
- Canada (2):
  - Toronto
  - Vancouver
- Germany (4):
  - Essen
  - Frankfurt am Main
  - Hamburg
  - München
- Italy (10):
  - Avellino
  - Benevento
  - Bologna
  - Padua
  - Parma
  - Pavia
  - Pisa
  - Reggio Emilia
  - Roma
  - Rozzano Milano

REFERENCES:
- [Derived] Santoro A, Rimassa L, Borbath I, Daniele B, Salvagni S, Van Laethem JL, Van Vlierberghe H, Trojan J, Kolligs FT, Weiss A, Miles S, Gasbarrini A, Lencioni M, Cicalese L, Sherman M, Gridelli C, Buggisch P, Gerken G, Schmid RM, Boni C, Personeni N, Hassoun Z, Abbadessa G, Schwartz B, Von Roemeling R, Lamar ME, Chen Y, Porta C. Tivantinib for second-line treatment of advanced hepatocellular carcinoma: a randomised, placebo-controlled phase 2 study. Lancet Oncol. 2013 Jan;14(1):55-63. doi: 10.1016/S1470-2045(12)70490-4. Epub 2012 Nov 20. PMID 23182627